CLINICAL TRIAL: NCT02408744
Title: Utility of Prolonged-release Pirfenidone in the Progression of Chronic Kidney Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Cell Therapy And Technology, S.a. De C.v. (Industry)
Responsible Party: Principal Investigator, Juan Armendáriz-Borunda, Head, Molecular Biology and Genomics Departament, CUCS, University of Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pirfenidona 001
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Fibrosis; Chronic Kidney Disease
Keywords: nephroprotection; pirfenidone; polymorphisms
MeSH Terms: conditions — Fibrosis; Renal Insufficiency, Chronic | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pirfenidone (Experimental): Pirfenidone 1200 mg in the form of prolonged-released tablets, orally administered two times a day (b.i.d.) to yield a daily dose of 2400 mg during three years.
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone was supplied orally in the form of prolonged-released tablets according with body surface area (m2 BS) of each patient. The target dosage of PFD was 1200 mg two times a day (b.i.d.) for a full dosage of 2400 mg daily during three years. Therapy was initiated at 600 mg b.i.d. and escalated to full dosage after 3 weeks when symptoms were controlled.
  Other Names: 5-methyl-1-phenyl-2-(1H)-pyridone

SUMMARY:
The aim of this study was to evaluate the impact in safety and efficacy of a new formulation of prolonged-released Pirfenidone in the progression of renal damage in patients with Chronic kidney Disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 10 and 40 years old with CKD
2. Diagnosis of CKD stage 1 to 4 according with KDIGO definition and classification
3. No glucocorticoids, cyclophasphamide, mycophenolate, or other immunosuppressive drugs for at least two months before starting PFD administration
4. Sign of consent forms

Exclusion Criteria:

1. Known intolerance to PFD
2. CKD stage V according with KDOQI classification
3. Post-transplant patients
4. History of peptic ulcer within six months
5. History of cerebrovascular disease within six months
6. Evidence of hepatic disease
7. Pregnancy or breast feeding
8. Malignancy

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the results of the use of Pirfenidone in the progression of renal damage in patients with Chronic Kidney Disease. | three years
  The progression of renal damage in patients with Chronic Kidney Disease was evaluated according to stages 1-4 of classification KDIGO.

SECONDARY OUTCOMES:
Effect of the use of Pirfenidone in renal function | Three years
  The renal function was monitored by cystatin C, reciprocal of serum creatinine and creatinine clearance collection of 24 hrs.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Armendariz-Borunda, Ph.D., Study Director — Head, Molecular Biology and Genomics Department, University of Guadalajara